CLINICAL TRIAL: NCT00958126
Title: A Phase II, Multicenter, Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Immunogenicity, Safety and Tolerability of CSL's 2009 H1N1 Influenza Vaccine (CSL425) in Healthy Adults Aged 18 Years and Older
Brief Title: A Clinical Trial of CSL's 2009 H1N1 Influenza Vaccine (CSL425) in Healthy Adults in the USA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-CAL-09-61
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2012-10-03 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CSL425 (7.5 mcg) (Experimental): 7.5 mcg of hemagglutinin antigen per dose. 0.25 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21
  Interventions: Biological: CSL425
- CSL425 (15 mcg) (Experimental): 15 mcg of hemagglutinin antigen per dose. 0.25 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21.
  Interventions: Biological: CSL425
- CSL425 (30 mcg) (Experimental): 30 mcg of hemagglutinin antigen per dose. 0.5 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21
  Interventions: Biological: CSL425
- Placebo (Placebo Comparator): Vaccine diluent. 0.5 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CSL425 — CSL's 2009 H1N1 Influenza Vaccine, thimerosal-free.
  Arms: CSL425 (7.5 mcg)
Biological: CSL425 — CSL's 2009 H1N1 Influenza Vaccine, thimerosal 0.01% (weight/volume).
  Arms: CSL425 (15 mcg); CSL425 (30 mcg)
Biological: Placebo — Vaccine diluent, thimerosal 0.01% (weight/volume).
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether CSL425 is a safe and effective vaccine for eliciting an immune response to H1N1 influenza in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and older, inclusive, at the time of providing informed consent.
* Females of child bearing potential (i.e., ovulating, pre-menopausal, not surgically sterile) must be abstinent or be willing to use a medically accepted contraceptive regimen for the duration of the study. Females of child bearing potential must return a negative urine pregnancy test result at enrolment and prior to each study vaccination.

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza virus vaccine or allergy to eggs, chicken protein, thimerosal, neomycin, polymyxin, or any components of the Study Vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1313 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Vaccines Clinical Development, Study Director — Seqirus
Locations (11):
- United States (11):
  - Study Site, Huntsville, Alabama
  - Study Site, San Diego, California
  - Study Site, Melbourne, Florida
  - Study Site, Peoria, Illinois
  - Study Site, South Bend, Indiana
  - Study Site, Metairie, Louisiana
  - Study Site, Baltimore, Maryland
  - Study Site, Rockville, Maryland
  - Study Site, Austin, Texas
  - Study Site, Fort Worth, Texas
  - Study Site, Salt Lake City, Utah

REFERENCES:
- [Result] Talaat KR, Greenberg ME, Lai MH, Hartel GF, Wichems CH, Rockman S, Jeanfreau RJ, Ghosh MR, Kabongo ML, Gittleson C, Karron RA. A single dose of unadjuvanted novel 2009 H1N1 vaccine is immunogenic and well tolerated in young and elderly adults. J Infect Dis. 2010 Nov 1;202(9):1327-37. doi: 10.1086/656601. PMID 20874515

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Adults: Vaccine diluent; Adults aged 18 to 64 years
- CSL425 (7.5 mcg), Adults: 7.5 mcg of hemagglutinin antigen per dose; Adults aged 18 to 64 years
- CSL425 (15 Mcg), Adults: 15 mcg of hemagglutinin antigen per dose; Adults aged 18 to 64 years
- CSL425 (30 Mcg), Adults: 30 mcg of hemagglutinin antigen per dose; Adults aged 18 to 64 years
- Placebo, Older Adults: Vaccine diluent; Older adults aged 65 years or older
- CSL425 (7.5 Mcg), Older Adults: 7.5 mcg of hemagglutinin antigen per dose; Older adults aged 65 years or older
- CSL425 (15 Mcg), Older Adults: 15 mcg of hemagglutinin antigen per dose; Older adults aged 65 years or older
- CSL425 (30 Mcg), Older Adults: 30 mcg of hemagglutinin antigen per dose; Older adults aged 65 years or older
Period: Overall Study
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Started | 49 | 205 | 201 | 203 | 50 | 203 | 200 | 202
Completed | 48 | 196 | 191 | 192 | 50 | 202 | 199 | 202
Not Completed | 1 | 9 | 10 | 11 | 0 | 1 | 1 | 0
Not completed — Serious Adverse Event | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Moved away from study area | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 5 | 9 | 8 | 0 | 0 | 0 | 0
Not completed — Sponsor/Investigator decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other Reason | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults | Total
Number analyzed (Participants) | 49 | 205 | 201 | 203 | 50 | 203 | 200 | 202 | 1313
Age, Customized [Number; unit: participants]
  >= 18 years to 64 years | 49 | 205 | 201 | 203 | 0 | 0 | 0 | 0 | 658
  >=65 years | 0 | 0 | 0 | 0 | 50 | 203 | 200 | 202 | 655
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 123 | 113 | 113 | 29 | 120 | 108 | 112 | 749
  Male | 18 | 82 | 88 | 90 | 21 | 83 | 92 | 90 | 564

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate 21 Days After the First Vaccination
Description: Seroconversion rate: the proportion of participants achieving seroconversion in hemagglutination inhibition (HI) antibody titer. Seroconversion is defined as participants with a baseline titer of less than 1:10 achieving a post-vaccination HI antibody titer of 1:40 or more; or participants with a baseline HI titer of 1:10 or more achieving a four-fold or greater increase in post-vaccination HI titer.
Time Frame: 21 days after the first vaccination
Population: The Evaluable Population (for the first vaccination) comprised all randomized participants who received the first study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Number analyzed (Participants) | 48 | 200 | 195 | 199 | 48 | 201 | 197 | 200
percentage of participants | 0 [0.0 to 7.4] | 82 [76.0 to 87.1] | 88.2 [82.8 to 92.4] | 94.5 [90.3 to 97.2] | 2.1 [0.1 to 11.1] | 51.2 [44.1 to 58.3] | 58.9 [51.7 to 65.8] | 73.0 [66.3 to 79.0]

2. Secondary Outcome: Frequency and Intensity of Solicited Adverse Events After the First Vaccination
Description: Grade 3 solicited adverse event (AE) definitions: Prevented normal daily activities; Size > 100 mm for injection site redness or induration/swelling; Temperature 102.2°F (39.0°C) or more for fevers.
Time Frame: During the 7 days after the first vaccination
Population: The Safety Population (first vaccination) comprised all randomized participants who received the first vaccination and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Number analyzed (Participants) | 49 | 204 | 201 | 203 | 50 | 203 | 200 | 202
percentage of participants
  Any local solicited adverse event | 22.4 [11.8 to 36.6] | 28.9 [22.8 to 35.7] | 35.8 [29.2 to 42.9] | 52.7 [45.6 to 59.7] | 4.0 | 13.3 | 23.5 | 21.8
  Any pain at injection site | 14.3 [5.9 to 27.2] | 14.7 [10.1 to 20.3] | 17.4 [12.4 to 23.4] | 31.0 [24.7 to 37.9] | 2.0 | 2.0 | 4.0 | 6.9
  Grade 3 pain at injection site | 0 | 0 | 0 | 0.5 | 0 | 0 | 0 | 0
  Any redness at injection site | 0 | 1.0 | 0.5 | 1.0 | 0 | 0.5 | 1.0 | 0
  Grade 3 redness at injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any swelling/induration at injection site | 0 | 3.9 | 2.5 | 3.9 | 0 | 2.0 | 3.0 | 2.5
  Grade 3 swelling/induration at injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any tenderness at injection site | 18.4 | 23.5 | 32.8 | 46.8 | 4.0 | 10.3 | 20.0 | 18.3
  Grade 3 tenderness at injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any bruising at injection site | 0 | 4.4 | 4.0 | 1.0 | 0 | 1.5 | 3.0 | 1.5
  Grade 3 bruising at injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any solicited systemic adverse event | 28.6 | 35.3 | 34.8 | 40.9 | 18.0 | 16.7 | 24.0 | 22.8
  Any headache | 16.3 | 19.6 | 21.4 | 27.1 | 8.0 | 9.4 | 10.5 | 10.4
  Grade 3 headache | 0 | 1.0 | 1.0 | 0 | 0 | 0.5 | 0 | 0.5
  Any malaise | 8.2 | 10.8 | 16.4 | 17.2 | 10.0 | 5.4 | 9.5 | 11.9
  Grade 3 malaise | 0 | 1.0 | 1.0 | 0 | 0 | 0 | 0 | 0
  Any myalgia | 4.1 | 14.7 | 15.9 | 17.7 | 8.0 | 8.9 | 13.0 | 13.4
  Grade 3 myalgia | 0 | 0.5 | 0.5 | 0 | 0 | 0 | 0 | 0
  Any nausea | 4.1 | 6.4 | 8.0 | 7.9 | 2.0 | 1.0 | 2.5 | 3.5
  Grade 3 nausea | 0 | 0.5 | 0 | 0.5 | 0 | 0 | 0 | 0
  Any chills | 2.0 | 3.9 | 5.0 | 5.4 | 0 | 0.5 | 1.0 | 3.0
  Grade 3 chills | 0 | 0.5 | 0.5 | 0 | 0 | 0 | 0 | 0
  Any vomiting | 0 | 2.9 | 1.0 | 1.0 | 0 | 0 | 0.5 | 0.5
  Grade 3 vomiting | 0 | 0.5 | 0 | 0 | 0 | 0 | 0 | 0
  Any fever | 2.0 | 3.4 | 3.0 | 3.4 | 0 | 0 | 0.5 | 0.5
  Grade 3 fever | 0 | 0.5 | 1.0 | 0.5 | 0 | 0 | 0 | 0

3. Secondary Outcome: Duration of Solicited Local Adverse Events After the First Vaccination
Time Frame: During the 7 days after the first vaccination, and day 7 - day 21 for ongoing AEs
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Number analyzed (Participants) | 49 | 204 | 201 | 203 | 50 | 203 | 200 | 202
days
  Pain at injection site | 1.14 (0.378) | 1.87 (2.705) | 1.71 (0.926) | 1.91 (1.237) | 1.00 (NA) — n = 1 | 1.75 (0.957) | 1.75 (0.886) | 1.27 (0.594)
  Redness at injection site | NA (NA) — n = 0 | 1.00 (0.000) | 1.00 (NA) — n = 1 | 2.50 (0.707) | NA (NA) — n = 0 | 1.00 (NA) — n = 1 | 1.00 (0.000) | NA (NA) — n = 0
  Swelling/induration at injection site | NA (NA) — n = 0 | 1.56 (0.726) | 1.2 (0.447) | 3.38 (2.615) | NA (NA) — n = 0 | 6.00 (10.00) | 1.5 (0.837) | 3.2 (4.382)
  Tenderness at injection site | 2.1 (1.912) | 2.04 (2.813) | 1.85 (0.966) | 1.90 (1.082) | 1.5 (0.707) | 1.27 (0.550) | 1.71 (0.955) | 1.65 (1.075)
  Bruising at injection site | NA (NA) — n = 0 | 3.00 (2.539) | 2.25 (1.669) | 2.00 (0.000) | NA (NA) — n = 0 | 8.00 (11.269) | 4.33 (2.503) | 1.20 (0.447)

4. Primary Outcome: Seroconversion Rate 21 Days After the Second Vaccination
Description: Seroconversion rate: the percentage of participants achieving seroconversion in HI antibody titer. Seroconversion is defined as participants with a pre-vaccination titer of less than 1:10 achieving a post-vaccination HI antibody titer of 1:40 or more; or participants with a pre-vaccination HI titer of 1:10 or more achieving a four-fold or greater increase in post-vaccination HI titer.
Time Frame: 21 days after the second vaccination
Population: The Evaluable Population (for the second vaccination) comprised all randomized participants who received the second study vaccine; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Number analyzed (Participants) | 48 | 196 | 191 | 193 | 48 | 200 | 196 | 198
percentage of participants | 6.3 [1.3 to 17.2] | 83.2 [77.2 to 88.1] | 91.1 [86.1 to 94.7] | 95.9 [92.0 to 98.2] | 8.3 [2.3 to 20.0] | 59.5 [52.3 to 66.4] | 67.3 [60.3 to 73.9] | 75.3 [68.6 to 81.1]

5. Primary Outcome: Percentage of Participants Achieving an Hemagglutination Inhibition (HI) Antibody Titer of 1:40 or More 21 Days After the First Vaccination
Time Frame: 21 days after the first vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Number analyzed (Participants) | 48 | 200 | 195 | 199 | 48 | 201 | 197 | 200
percentage of participants | 22.9 [12.0 to 37.3] | 97.0 [93.6 to 98.9] | 96.4 [92.7 to 98.5] | 99.5 [97.2 to 100.0] | 39.6 [25.8 to 54.7] | 92.0 [87.4 to 95.4] | 90.9 [85.9 to 94.5] | 94.0 [89.8 to 96.9]

6. Primary Outcome: Percentage of Participants Achieving an HI Antibody Titer of 1:40 or More 21 Days After the Second Vaccination
Time Frame: 21 days after the second vaccination
Population: The Evaluable Population (for the second vaccination) comprised all randomized participants who received the second study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Number analyzed (Participants) | 48 | 196 | 191 | 193 | 48 | 200 | 196 | 198
percentage of participants | 29.2 [17.0 to 44.1] | 98.5 [95.6 to 99.7] | 99.5 [97.1 to 100.0] | 99.5 [97.1 to 100.0] | 35.4 [22.2 to 50.5] | 96.0 [92.3 to 98.3] | 93.4 [88.9 to 96.4] | 94.9 [90.9 to 97.6]

7. Secondary Outcome: Incidence of Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESI) and New Onset of Chronic Illness (NOCI)
Description: A NOCI was defined as the diagnosis of a new medical condition that was chronic in nature, including those potentially controllable by medication (eg, diabetes, asthma).
Time Frame: Up to 180 days after the last vaccination
Population: The Safety Population comprised all randomized participants who received at least one dose of study vaccine and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Number analyzed (Participants) | 49 | 204 | 201 | 203 | 50 | 203 | 200 | 202
percentage of participants
  Percentage of participants with at least one SAE | 0 | 2.9 | 2.0 | 1.5 | 6.0 | 4.4 | 3.0 | 4.5
  Percentage of participants with related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Percentage of participants with at least one AESI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Percentage of participants with related AESI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Percentage of participants with at least one NOCI | 4.1 | 0.5 | 0.5 | 0.5 | 2.0 | 1.0 | 2.5 | 2.0
  Percentage of participants with related NOCI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Frequency and Intensity of Unsolicited Adverse Events (UAE) After the First or Second Vaccination
Description: Unsolicited adverse event (UAE) grading:
  Grade 1 (mild): Symptoms were easily tolerated and did not interfere with daily activities.
  Grade 2 (moderate): Enough discomfort to cause some interference with daily activities.
  Grade 3 (severe): Symptoms that prevented normal, everyday activities.
Time Frame: Day 0 to Day 20 after each vaccination; up to Day 180 after the last vaccination for SAEs, AESI and NOCI
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Groups:
- Placebo, Age Cohorts Combined: Vaccine diluent
- CSL425 (7.5 mcg), Age Cohorts Combined: 7.5 mcg of hemagglutinin antigen per dose
- CSL425 (15 Mcg), Age Cohorts Combined: 15 mcg of hemagglutinin antigen per dose
- CSL425 (30 Mcg), Age Cohorts Combined: 30 mcg of hemagglutinin antigen per dose
Arm/Group | Placebo, Age Cohorts Combined | CSL425 (7.5 mcg), Age Cohorts Combined | CSL425 (15 Mcg), Age Cohorts Combined | CSL425 (30 Mcg), Age Cohorts Combined
Number analyzed (Participants) | 99 | 407 | 401 | 405
percentage of participants
  Percentage of participants with at least one UAE | 27.3 | 27.5 | 30.2 | 27.9
  Percentage of participants reporting Grade 1 UAE | 7.1 | 12.8 | 10.0 | 12.8
  Percentage of participants reporting Grade 2 UAE | 15.2 | 8.8 | 14.0 | 10.4
  Percentage of participants reporting Grade 3 UAE | 5.1 | 5.9 | 6.2 | 4.7

ADVERSE EVENTS:
Time Frame: For SAEs: up to 180 days after the last vaccination. For unsolicited adverse events: 21 days after the first study vaccination, up to 180 days after the the last vaccination (for AESI and NOCI).
Description: Serious Adverse Events were collected from Day 0 to 180 days after the last vaccination.
  The other adverse events presented are unsolicited adverse events from Day 0 to Day 20 days after the first study vaccination, AESI and NOCI from Day 0 to 180 days after the last vaccination.
Arm/Group | Placebo, Adults | CSL425 (7.5 mcg), Adults | CSL425 (15 Mcg), Adults | CSL425 (30 Mcg), Adults | Placebo, Older Adults | CSL425 (7.5 Mcg), Older Adults | CSL425 (15 Mcg), Older Adults | CSL425 (30 Mcg), Older Adults
Serious Adverse Events (participants affected / at risk) | 0/49 | 6/204 | 4/201 | 3/203 | 3/50 | 9/203 | 6/200 | 9/202
Other Adverse Events (participants affected / at risk) | 12/49 | 27/204 | 25/201 | 27/203 | 5/50 | 20/203 | 23/200 | 18/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Adults (N=49) | CSL425 (7.5 mcg), Adults (N=204) | CSL425 (15 Mcg), Adults (N=201) | CSL425 (30 Mcg), Adults (N=203) | Placebo, Older Adults (N=50) | CSL425 (7.5 Mcg), Older Adults (N=203) | CSL425 (15 Mcg), Older Adults (N=200) | CSL425 (30 Mcg), Older Adults (N=202)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral myocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung metastatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo, Adults (N=49) | CSL425 (7.5 mcg), Adults (N=204) | CSL425 (15 Mcg), Adults (N=201) | CSL425 (30 Mcg), Adults (N=203) | Placebo, Older Adults (N=50) | CSL425 (7.5 Mcg), Older Adults (N=203) | CSL425 (15 Mcg), Older Adults (N=200) | CSL425 (30 Mcg), Older Adults (N=202)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 8 (8) | 5 (7) | 4 (4) | 0 (0) | 7 (8) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 8 (8) | 8 (8) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 7 (7) | 9 (9) | 0 (0) | 3 (4) | 1 (1) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 5 (5) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (2) | 2 (3) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0/0 (0) | 0 (0) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.